CLINICAL TRIAL: NCT04351776
Title: Functional Outcome Response to Engaging Virtual Reality in Pediatric Patients: a Randomized Clinical Trials
Brief Title: Virtual Reality and Pain
Acronym: FOREVR Peds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-1090
Record Dates: First submitted 2020-04-03; First posted 2020-04-17 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Pain, Postoperative; Pain; Anxiety Postoperative
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Intervention Model Description: 90 participants assigned to one of three groups (30 participants for each group). VR- Biofeedback, VR-Distraction, 360 Video
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR-Biofeedback (Other)
  Interventions: Other: VR-Biofeedback
- VR-Distraction (Other)
  Interventions: Other: VR-Distraction
- 360 Video (Other)
  Interventions: Other: 360 Video

INTERVENTIONS:
Other: VR-Biofeedback — Participants will be instructed to use the Mindful Aurora application
  Arms: VR-Biofeedback
Other: VR-Distraction — Participants will be instructed to use one of three applications
  Arms: VR-Distraction
Other: 360 Video — Participants will be instructed which video to view
  Arms: 360 Video

SUMMARY:
Determine the impact of VR-Biofeedback, VR-distraction, and 360 video on pain and medication utilization in patients undergoing surgery; determine the role of anxiety and pain catastrophizing on changes in pain following VR-BF in patients undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ages 8 - 18 years
* Able to read, understand and speak English
* Patients in the immediate postoperative period with significant pain being followed by the Acute Pain Service

Exclusion Criteria:

* Outside the age range (< 8 or > 18 years)
* History of developmental delays, uncontrolled psychiatric conditions, or neurological conditions (especially epilepsy and/or significant motion sickness/nausea/vomiting)
* History of vertigo, dizziness, and/or seizure disorder
* Conditions that would preclude the application of the VR headset, such as surgeries of the head and neck

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Effect of VR-biofeedback on pain | Postoperatively 24 - 90 hours.
  Pain scores will be collected. Pain will be rated using the numerical rating scale. Participant will rate their pain from 0 - 10. 0 meaning no pain and 10 being the worst pain imaginable.
Effect of VR-distraction on pain | Postoperatively 24 - 90 hours.
  Pain scores will be collected. Pain will be rated using the numerical rating scale. Participant will rate their pain from 0 - 10. 0 meaning no pain and 10 being the worst pain imaginable.
Effect of 360 video on pain | Postoperatively 24 - 90 hours.
  Pain scores will be collected. Pain will be rated using the numerical rating scale. Participant will rate their pain from 0 - 10. 0 meaning no pain and 10 being the worst pain imaginable.

SECONDARY OUTCOMES:
Effect of VR-biofeedback on anxiety | Before 10 minute VR session.
  Anxiety scores will be collected. Anxiety will be rated using a visual analog scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety.
Effect of VR-biofeedback on anxiety | After 10 minute VR session. Anxiety will be rated using a visual analog scale.
  Anxiety scores will be collected. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety
Effect of VR-biofeedback on medication use | Duration of hospital stay up to 30 days after discharge
  Medications used will be collected
Effect of VR-distraction on anxiety | Before 10 minute VR session.
  Anxiety scores will be collected. Anxiety will be rated using a visual analog scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety
Effect of VR-distraction on anxiety | After 10 minute VR session.
  Anxiety scores will be collected. Anxiety will be rated using a visual analog scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety
Effect of VR-distraction on medication use | Duration of hospital stay up to 30 days after discharge
  Medications used will be collected
Effect of 360 video on anxiety | Before 10 minute VR session.
  Anxiety scores will be collected. Anxiety will be rated using a visual analog scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety
Effect of 360 video on anxiety | After 10 minute VR session.
  Anxiety scores will be collected. Anxiety will be rated using a visual analog scale. Anxiety will be rated from 0 - 10. 0 meaning no anxiety 10 being severe anxiety
Effect of 360 video on medication use | Duration of hospital stay up to 30 days after discharge
  Medications used will be collected
Role of anxiety on changes in pain | One time prior to study visit
  Participants will complete a questionnaire regarding anxiety
Role of pain catastrophizing | One time prior to study visit
  Participants will complete a questionnaire regarding pain

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Walter, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
This information will be made available upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available upon publication. All data will be deidentified.

REFERENCES:
- [Derived] Olbrecht VA, Williams SE, O'Conor KT, Boehmer CO, Marchant GW, Glynn SM, Geisler KJ, Ding L, Yang G, King CD. Guided relaxation-based virtual reality versus distraction-based virtual reality or passive control for postoperative pain management in children and adolescents undergoing Nuss repair of pectus excavatum: protocol for a prospective, randomised, controlled trial (FOREVR Peds trial). BMJ Open. 2020 Dec 30;10(12):e040295. doi: 10.1136/bmjopen-2020-040295. PMID 33380482